CLINICAL TRIAL: NCT05665049
Title: Social Transfers for Exclusive Breastfeeding: A Pilot Program in Lao People's Democratic Republic (Lao PDR)
Brief Title: Social Transfers for Exclusive Breastfeeding
Acronym: STEB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Lao Tropical and Public Health Institute (Lao TPHI) (Unknown); University of Basel (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: steb1
Record Dates: First submitted 2022-10-21; First posted 2022-12-27 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Feeding, Exclusive; Breastfeeding; Development, Child; Development, Infant
Keywords: breastfeeding; early childhood development; social transfer; cash transfer
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Only educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided.
- Intervention Group 1 - Non-Conditional Social Transfer (Experimental): Educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided. At the baseline visit, participants are told that at the 6-month visit, they will receive a gift of their choice - which is meant to show our appreciation and support for their efforts in breastfeeding.
  Interventions: Behavioral: Social Transfer
- Intervention Group 2 - Conditional Social Transfer (Experimental): Educational materials focused on the benefits of exclusive breastfeeding and the current international recommendations are provided. At the baseline visit, participants are told that at the 6-month visit, they will receive a gift of their choice if they are still exclusively breastfeeding.
  Interventions: Behavioral: Social Transfer

INTERVENTIONS:
Behavioral: Social Transfer — Social transfers are defined as a cash or in-kind transfer. Using results from a qualitative study, we identified the following culturally grounded social transfer options that is responsive to the identified needs of new mothers. Based on the monthly Lao PDR minimum wage and an estimated 15 full working days needed to exclusively breastfeed over a 6-month period, a social transfer of approximately $75 would fairly subsidize women's breastfeeding efforts. Therefore all social transfer options equate to approximately 75 USD. The options include: diapers, child developmental toys, cash, or a combination of these.
  Arms: Intervention Group 1 - Non-Conditional Social Transfer; Intervention Group 2 - Conditional Social Transfer

SUMMARY:
The goal of this study is to assess the effectiveness of social transfers on exclusive breastfeeding rates in Lao PDR. The main questions it aims to answer are:

1. Are social transfers effective at increasing exclusive breastfeeding rates at 6-months
2. Are social transfers cost-effective
3. What are the long-term impacts of social transfers for breastfeeding on child development

Participants will be randomly assigned to one of three groups: 1) control, no social transfer 2) non-conditional social transfer at 6-months postpartum, and 3) conditional social transfer at six months postpartum; conditional upon the mothers exclusive breastfeeding status.

All participants receive education about the benefits of exclusive breastfeeding and current international recommendations.

Researchers will compare the intervention groups to the control group to see if social transfers are effective at increasing exclusive breastfeeding rates at six months postpartum.

ELIGIBILITY:
Inclusion criteria:

* Given birth in the last four weeks
* Exclusively breastfeeding at time of recruitment
* Lives in Vientiane in one of the following districts: Chanthabury, Sikhottabong, Sangthong, or Parkngum and is included in the VITERBI cohort

Exclusion criteria:

* Plans to move permanently outside study area
* Has a medical, intellectual or psychological disability
* Contraindication for breastfeeding
* Preterm births
* Children born with < 2500 grams

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Exclusive Breastfeeding at 6-Months Postpartum | 6 Months Postpartum
  The primary endpoint is the proportion of women exclusively breastfeeding at 6-months postpartum assessed using a questionnaire. Exclusive breastfeeding is defined as receipt of only human milk - which is consistent with the World Health Organization guidelines. At six months postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the exclusive breastfeeding status.

SECONDARY OUTCOMES:
Anthropometric Measurements | 1 month, 6 months, 1 year, 2 years, 3 years
  Infants will be measured for length, weight, head circumference, skinfold thickness. Height was measured in centimeters by using a Height Measuring Device, stadiometer, 20-205cm. Weight was measured in kilograms by a mobile weighing scale. Skin fold measurements were collected using a skin fold caliper. Head, waist, and hip measurements and MUAC were measured using non-stretchable measuring tape. All measurements will be analyzed as age standardized z-scores.
Mother and Child Anemia Levels | 1 month, 6 months, 1 year, 2 years, 3 years
  We will assess the mother and child anemia levels. The HemoCue Hb 301 will be used to give an instant measurement of the Haemoglobin (Hb) level of the patient. Capillary blood will be collected through a finger prick. Blood samples drawn for the haemoglobin assessment will be discarded after the test. Iron levels will be analyzed as a continuous outcome.
Early Childhood Development | 2 years
  When the child is two years of age, a comprehensive end line assessment will be conducted to evaluate early childhood development indicators (e.g. The Global Scale for Early Development (GSED). This indicator will be normalized to a mean of 0 and SD of 1 to facilitate interpretation of estimated group differences.
Early Childhood Development | 3 years
  When the child is three years of age, the IDELA will assess children's cognitive, social and language skills, and lifelong capacity for learning. This indicator will be normalized to a mean of 0 and SD of 1 to facilitate interpretation of estimated group differences.
Complementary Breastfeeding Duration | 6 months, 1 year, 2 years
  The proportion of women complementary breastfeeding at 6-months, 1-year, and 2-years postpartum assessed using a questionnaire. Complementary breastfeeding is defined as receipt of human milk in combination with complementary foods and liquid. At each time point postpartum, mothers are asked if they are still currently breastfeeding. If they answer yes, a follow-up question on if they provided any other liquids, solids, or supplements to their child to determine the complementary breastfeeding status.

CONTACTS AND LOCATIONS:
Overall Officials: Jordyn T Wallenborn, PhD, MPH, Principal Investigator — Swiss Tropical and Public Health Institute, University of Basel
Locations (1):
- Lao Tropical and Public Health Institute (Lao TPHI), Vientiane, Laos

REFERENCES:
- [Derived] Wallenborn JT, Sonephet S, Sayasone S, Siengsounthone L, Kounnavong S, Fink G. Conditional and Unconditional Social Transfers, Early-Life Nutrition, and Child Growth: A Randomized Clinical Trial. JAMA Pediatr. 2025 Feb 1;179(2):129-136. doi: 10.1001/jamapediatrics.2024.5079. PMID 39680397
- [Derived] Sonephet S, Kounnavong S, Zinsstag L, Vonaesch P, Sayasone S, Siengsounthone L, Odermatt P, Fink G, Wallenborn JT. Social Transfers for Exclusive Breastfeeding (STEB) Intervention in Lao People's Democratic Republic: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 May 3;13:e54768. doi: 10.2196/54768. PMID 38700928